CLINICAL TRIAL: NCT03939884
Title: MuscleCare™ Pain Relief Therapy vs. Voltaren® in the Relief of Trapezius Trigger Point Musculoskeletal Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Active and Innovative Inc. (Other)
Responsible Party: Principal Investigator, Jack Goodman, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MuscleCare_Voltaren
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Pain
Keywords: Analgesia; Myofascial Pain; MuscleCare; Voltaren; NSAID
MeSH Terms: conditions — Pain; Agnosia | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Professional Therapy Muscle Care™ roll-on with MSM (Experimental)
  Interventions: Drug: MuscleCare Topical Product
- Professional Therapy Muscle Care™ roll-on without MSM (Experimental)
  Interventions: Drug: MuscleCare Topical Product
- Professional Therapy Muscle Care™ Ointment with MSM (Experimental)
  Interventions: Drug: MuscleCare Topical Product
- Professional Therapy Muscle Care™ Ointment without MSM (Experimental)
  Interventions: Drug: MuscleCare Topical Product
- Voltaren Emulgel (Active Comparator)
  Interventions: Drug: Voltaren Topical
- Non-medicinal Placebo (Placebo Comparator)
  Interventions: Drug: Nivea, Topical Cream

INTERVENTIONS:
Drug: MuscleCare Topical Product — Application of the product will be applied with six circular applications over the trigger point and left to rest for 7 minutes.
  Arms: Professional Therapy Muscle Care™ Ointment with MSM; Professional Therapy Muscle Care™ Ointment without MSM; Professional Therapy Muscle Care™ roll-on with MSM; Professional Therapy Muscle Care™ roll-on without MSM
Drug: Voltaren Topical — Application of the product will be applied with six circular applications over the trigger point and left to rest for 7 minutes.
  Arms: Voltaren Emulgel
Drug: Nivea, Topical Cream — Application of the product will be applied with six circular applications over the trigger point and left to rest for 7 minutes.
  Arms: Non-medicinal Placebo

SUMMARY:
To determine the difference in efficacy of an all natural topical analgesic (MuscleCare) to a product containing the non-steroidal anti-inflammatory drug diclofenac (Voltaren) on trapezius trigger point pain.

DETAILED DESCRIPTION:
Myofascial pain syndromes (MPS) are common in Western society. Vernon and Schneider note that MPS is thought to be the leading diagnosis among pain management specialists and the leading diagnosis in pain patients reporting to general practitioners. MPS can be viewed as a regional pain syndrome such as, neck, low back and upper quadrant pain syndromes. MPS can also be found focally in discrete painful sites known as Myofascial Trigger Points (MTP). Locations of MTP's have been characterized on clinical grounds throughout the musculoskeletal system, starting with the seminal work of Travell and Simons. MTP's have been described as active (clinically active with pain referral upon palpation) or latent (not clinically active, but tender on manual palpation). The presence of associated features such as "local twitch sign" and palpable taut bands is thought to confirm the presence of an active MTP, while latent TP's may not present with the classic features.

Numerous treatments are currently available for MPS and MTP's. Several systematic reviews have recently been published on a variety of treatments, including pharmacologic agents, physical agents, complementary and alternative therapies. One commonly used therapy is the application of topical agents to relieve pain. These agents can be classified as pharmacologic or non-pharmacologic. The former category includes non-steroidal anti-inflammatory agents (such as ketoprofen), opioid agents, classical analgesic agents (such as lidocaine), novel analgesic agents such as capsaicin and rubefascient agents (containing salicylates or nicotinamides). Non-pharmacologic agents generally fall into the complementary and alternative medicine (CAM) category for MPS and MTP treatments. They may contain putative analgesic agents or counterirritant agents and they may exert cold, hot or neutral effects.

The literature on myofascial trigger points and non-pharmacologic topical agents is sparse with no randomized clinical trials found to date. Several studies have investigated the effect of such topicals in the treatment of osteoarthritis, particularly of the knee. However, there appears to be a lack of studies investigating the effects of topicas for the treatment of MPS or MTP. A randomized, placebo-blinded clinical trial of non-pharmacological topical analgesics is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years old

Exclusion Criteria:

* acute pain presentation preventing comfortable participation, absence of a palpable tender spot in the right upper trapezius region (this feature will be identified by manual palpation by a neutral assessor prior to enrollment), any history of allergic reaction to previous use of any analgesic topicals, any disorder of the skin over the right trapezius area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Baseline (Pre product application) and 7 minutes post product application
  Change in pressure pain threshold by pressure algometry over the target MTP in the upper trapezius and will be reported in kg/sq.cm

CONTACTS AND LOCATIONS:
Overall Officials: Jack Goodman, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Avrahami D, Hammond A, Higgins C, Vernon H. A randomized, placebo-controlled double-blinded comparative clinical study of five over-the-counter non-pharmacological topical analgesics for myofascial pain: single session findings. Chiropr Man Therap. 2012 Mar 21;20:7. doi: 10.1186/2045-709X-20-7. PMID 22436614